CLINICAL TRIAL: NCT07198477
Title: Sleep Disturbances and Their Association With Serum Magnesium Level in Patients With Major Depressive Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Aref Fouad, resident at the Neuropsychiatry department, Assiut University
Other Study IDs: Mg levels in major depression
Record Dates: First submitted 2025-09-29; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder; Sleep Disturbances
Keywords: sleep disturbances
MeSH Terms: conditions — Depressive Disorder; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with major depressive disorder: The study sample will include 90 psychiatric patients recruited from the outpatient and inpatient clinics of Assiut University Hospital, representing males and females aged 18-60 years. All participants will have a confirmed diagnosis of major depressive disorder based on clinical criteria and will be evaluated using standardized psychiatric assessment tools.

SUMMARY:
This cross-sectional study investigates the relationship between serum magnesium levels and the presence of sleep disturbances among patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Major depressive disorder is a highly prevalent psychiatric condition often accompanied by disabling sleep disturbances, including insomnia and hypersomnia. Evidence suggests that magnesium, a vital trace element involved in neurotransmission, stress response, and circadian regulation, may play a crucial role in both mood and sleep. Low serum magnesium levels have been linked to increased depressive symptom severity and disturbed sleep quality. This study seeks to explore whether hypomagnesemia can serve as a biological contributor to sleep dysfunction in MDD. By employing the Beck Depression Inventory-II (BDI-II) and the Pittsburgh Sleep Quality Index (PSQI), as well as laboratory measurement of serum magnesium levels, the study aims to determine whether lower magnesium is significantly associated with greater depressive burden and poor sleep outcomes. The findings may help validate magnesium as a biomarker for early screening and risk stratification in psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of major depressive disorder

age 18 years and older

Ability to complete questionnaires (BDI-II and PSQI; validated Arabic versions)

Willing to participate and provide informed consent

Exclusion Criteria:

* hronic renal failure or metabolic disorders affecting magnesium balance

Current use of medications known to significantly interfere with serum magnesium (e.g., long-term diuretics, proton pump inhibitors) unless stable and documented

Presence of other comorbid psychiatric disorders

Cognitive impairment or language difficulties preventing questionnaire completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will include 90 psychiatric patients recruited from the outpatient and inpatient clinics of Assiut University Hospital, representing males and females aged 18-60 years. All participants will have a confirmed diagnosis of major depressive disorder based on clinical criteria and will be evaluated using standardized psychiatric assessment tools. Exclusion criteria were designed to rule out metabolic comorbidities, chronic renal conditions, and medication effects that may confound serum magnesium interpretation. Patients unable to complete questionnaires due to cognitive or language difficulties, as well as those with other psychiatric disorders, will also be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
change in the level of serum magnesium level | Baseline
  Serum magnesium concentration (mmol/L) measured by atomic absorption spectrophotometry for the patients.